CLINICAL TRIAL: NCT05064813
Title: Elucidating Neural Mechanisms and Sex Differences in Response to Mindfulness Based Stress Reduction in Generalized Anxiety Disorder
Brief Title: MBSR Mechanisms in GAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-00454
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction Group (Experimental): 8 weeks of Mindfulness Based Stress Reduction Group (MBSR).
  Interventions: Behavioral: Mindfulness Based Stress Reduction MBSR Intervention
- Stress Education Group (Active Comparator): 8 weeks of Stress Education Group (SE).
  Interventions: Behavioral: Stress Education Control Condition (SE)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction MBSR Intervention — MBSR is an 8-week group-based course developed by Jon Kabat-Zinn (1990) and colleagues at the University of Massachusetts' Center for Mindfulness. Weekly 2.5 hour long classes are given once a week, as well as one day-long weekend class. The classes instruct participants in the theory and practice of several forms of mindfulness meditation, breathing awareness, and mindfulness stretching exercises. Teaching of the theory of mindfulness and experiential practice are both utilized during weekly classes and at-home CD-guided practice sessions.
  Arms: Mindfulness Based Stress Reduction Group
Behavioral: Stress Education Control Condition (SE) — Stress Education (SE) was designed to provide an active comparator condition that does not include overlapping active components of mindfulness meditation with MBSR. It will also be delivered over 8-weekly, in-person, 2.5 hour group sessions of the same size (n=4 to 6). In SE, participants receive extensive information about stress and health, but will not receive any MBSR or other mind-body training. Instead, stress relevant psycho-educational information will be taught.
  Arms: Stress Education Group

SUMMARY:
The purpose of this study is to understand the neural mechanisms that drive response to MBSR compared to stress education in patients with generalized anxiety disorder (GAD), and to examine the degree to which sex differences in MBSR response are explained by sex differences in these mechanisms. A total of 150 eligible participants with a primary diagnosis of GAD will be randomized to either an 8-week group MBSR or stress education program. The study will include preliminary screening, experimental visits, including fMRI, group intervention visits, and assessments at baseline, endpoint, and 3-month follow-up.

DETAILED DESCRIPTION:
Mindfulness-Based Stress Reduction (MBSR) has demonstrated efficacy for Generalized Anxiety Disorder (GAD), yet there remains a major knowledge gap about its neural mechanisms.

This study will examine functional activation of brain regions associated with the fear extinction network (ventromedial prefrontal cortex (vmPFC), hippocampus, and amygdala) as a specific probe of the 'instinctual' type of emotion regulation as well as large-scale functional connectivity as a marker of neural plasticity changes. Sex differences in MBSR-induced neural changes and their relationship to sex differences in clinical GAD response will be examined. Finally, a novel statistical approach will be used to explore whether baseline neural measures can predict neural changes and clinical symptom reduction to identify likely MBSR responders.

The unique combination of a focus on GAD, an anxiety condition with established emotion regulation difficulties implicating target neural circuits, previously demonstrated MBSR efficacy, and sex differences with rigorous fMRI behavioral probes with novel analytic approaches ought to provide major new insights about MBSR versus stress education mechanisms and sex considerations, moving towards precision medicine that could guide future treatment development research.

Eligible participants with Generalized Anxiety Disorder will be 2:1 randomized to group intervention with MBSR or stress education classes. They will participate for 13-14 weeks plus one 3 month follow up assessment (23-24 weeks from screening). Full participation includes screening, baseline, endpoint and 3 month follow up assessments, two sets of experimental days 12 weeks apart which include fMRI scans, and 8 weeks of the assigned group intervention (either MBSR or stress education).

ELIGIBILITY:
Inclusion Criteria:

* Male or pre-menopausal female outpatients aged 18 to 50 years of age
* A primary mental health complaint (designated by the patient as the most important source of current distress and confirmed on structured clinical interview for DSM-5 diagnoses by a certified clinical evaluator) of Generalized Anxiety Disorder (GAD), as defined by DSM-5 criteria.
* Overall clinical anxiety severity of at least mild as defined by a CGI-S of at least 3.
* Willingness and ability to participate in the informed consent process and comply with the requirements of the study protocol.

Exclusion Criteria:

* A lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders; obsessive-compulsive disorder or an eating disorder in the past 12 months; neurocognitive disorders, intellectual disabilities, communication disorders or other cognitive dysfunction that could interfere with capacity to engage in therapy or complete study procedures; substance or alcohol use disorder (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
* Patients with significant suicidal ideation (assessed by CSSR-S SI score greater than 2) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Patients must be free of concurrent benzodiazepine, antipsychotic, and stimulant medication for at least 4 weeks prior to initiation of randomized treatment. Other psychiatric medications such as antidepressants that have been stable for at least 4 weeks prior to randomization will be permitted.
* Inability to understand study procedures or informed consent process, or significant personality dysfunction likely to interfere with study participation (assessed during the clinical interview) or inability to comply with study procedures (such as planned extended travel) assessed on clinical interview
* Serious current unstable medical illness, or a condition for which hospitalization may be likely within the next year as assessed by medical history and physical exam. If any questions about medical safety emerge, consent will be formally obtained to contact patient's PCP in order to determine whether any medical concerns making participation unsafe or not feasible (such as need for extended inpatient care) are present; MBSR and SE, however, do not require intensive exercise capacity or mobility.
* Pregnant women (to be ruled out by urine ß-HCG) and women of childbearing potential who are not using medically accepted forms of contraception (such as IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
* Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of GAD or with any mindfulness and/or meditation component is excluded. Prohibited psychotherapy includes CBT, DBT, ACT, mindfulness based approaches, or psychodynamic therapy focusing on exploring specific, dynamic causes of the GAD symptomatology and providing management skills. General supportive therapy initiated greater than 3 months prior is acceptable.
* Individuals who have completed a course of MBSR or an equivalent meditation training or who have an ongoing regular meditation practice in the past 2 years.
* Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
* Contraindications for MRI including metal implants, surgical clips, probability of metal fragments, or braces that are prohibited due to severe risk of injury.
* Left handed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-post changes in fMRI measures of functional activation in the fear extinction network during fear extinction learning | Experimental Days 1 & 2 (Visit 2 & 3) and Experimental Days 3 & 4 (Visit 9 & 10)
  The primary clinical outcome measure will be treatment response. This is measured by The Clinical Global Impression-Improvement (CGI-I) scale is a single clinician-reported item that assesses how much the patient's illness has improved or worsened relative to baseline and is rated as 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse,) 6 (much worse), or 7 (very much worse). The CGI-I scale is widely used and well validated, and is sensitive to changes in neuropsychiatric symptoms.
Pre-post changes in fMRI measures of functional activation in the whole brain neural connectivity during fear extinction learning | Experimental Days 1 & 2 (Visit 2 & 3) and Experimental Days 3 & 4 (Visit 9 & 10)
  The primary clinical outcome measure will be treatment response. This is measured by The Clinical Global Impression-Improvement (CGI-I) scale is a single clinician-reported item that assesses how much the patient's illness has improved or worsened relative to baseline and is rated as 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse,) 6 (much worse), or 7 (very much worse). The CGI-I scale is widely used and well validated, and is sensitive to changes in neuropsychiatric symptoms.

SECONDARY OUTCOMES:
Change in Skin Conductance Response (SCR). | Experimental Days 1 & 2 (Visit 2 & 3) and Experimental Days 3 & 4 (Visit 9 & 10)
  SCR will be computed for each trial by subtracting the mean SCR during the last seconds of context presentation from the maximal skin conductance response reached during CS presentation during the fear conditioning and extinction paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Simon, MD, Principal Investigator — NYU Langone Health; Candace Raio, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The primary cleaned deidentified dataset 12 months after database lock or primary publication or whatever comes first
Supporting Information: Study Protocol, SAP
Time Frame: This data will be made available within twelve months of database lock or following publication of primary manuscript, whichever occurs first.
Access Criteria: Anyone who wishes to access the data. Any purpose. A de-identified dataset can be readily shared without the need of a Data Use Agreement (DUA) and facilitates book-keeping, making it the preferred data sharing plan. NYU SoM is committed to creating limited access public use datasets in accordance with NIH specifications. All study data will be made available via a data archive accessible through a public website hosted and maintained by NYU SoM. Web archived data may also be available as downloadable content, facilitating access to the research data.